CLINICAL TRIAL: NCT06726239
Title: The Effect of Progressive Relaxation Exercises Applied Before Mobilization on Pain, Anxiety and Physiological Parameters in Patients With Coronary Artery Bypass Graft Surgery
Brief Title: Progressive Relaxation Exercises Before Mobilization:Effects on Pain, Anxiety and Physiologic Parameters CABG Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tugce Bozkurt Elmas, PhD Candidate in Surgical Nursing, Istanbul University-Cerrahpasa, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1308
Record Dates: First submitted 2024-12-02; First posted 2024-12-10 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Pain; Anxiety; Physiological Parameter; Mobilization; Coronary Artery Bypass Graft Surgery (CABG); PROGRESSIVE MUSCLE RELAXATION EXERCISES
Keywords: coronary artery bypass graft surgery; pain; Anxiety; progressive relaxation exercise; physiological parameter
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: experiment-control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): In the preoperative period, patients in the control group completed the Patient Demographic Information Form and the Trait Anxiety Inventory. Patients were preoperatively informed about wearing a smart bracelet on postoperative days 1 and 2 to track step count and walking distance. Physiological parameters, state anxiety, and pain levels (Short-Form McGill Pain Questionnaire) were evaluated at pre-test, 30 minutes later, and 15 minutes after mobilization. Additionally, pain intensity was assessed immediately after mobilization. On postoperative days 1 and 2, all assessments were conducted twice daily. The frequency of analgesic administration was also monitored.
- Experimental (Experimental): In the preoperative period, patients completed the Patient Demographic Information Form and the Trait Anxiety Inventory. Patients were preoperatively informed about wearing a smart bracelet on postoperative days 1 and 2 to track step count and walking distance. Furthermore, patients in the intervention group received video-assisted training on diaphragmatic breathing and progressive muscle relaxation (PMR) exercises.
  In the intervention group, PMR was performed twice a day on postoperative days 1 and 2. Physiological parameters, state anxiety, and pain levels (Short-Form McGill Pain Questionnaire) were measured at pre-test, 5 minutes after each PMR session, and 15 minutes after mobilization. Additionally, pain intensity was assessed immediately after mobilization. The frequency of analgesic administration was also monitored.
  Interventions: Other: Progressive relaxation exercises

INTERVENTIONS:
Other: Progressive relaxation exercises — The aim of relaxation exercises is to help individuals recognize the difference between tension and relaxation and to enable them to relax in situations of stress. These exercises are performed with light background music and verbal instructions, allowing patients to mentally focus on the process. The progressive relaxation technique involves the voluntary contraction and subsequent relaxation of muscle groups, typically starting from the hands and progressing to the feet, with each muscle group activated in sequence. During the exercise, the instructions and steps from the 'Relaxation Exercises' CD published by the Turkish Psychologists Association will be followed.
  Arms: Experimental

SUMMARY:
This study is planned as a randomized controlled experimental study to determine the effect of progressive relaxation exercises applied before mobilization on pain, anxiety and physiological parameters in patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled experimental study to determine the effect of progressive relaxation exercises on pain, anxiety and physiological parameters before mobilization in patients undergoing coronary artery bypass graft (CABG) surgery. Ethics committee and institutional approval were obtained before starting the study. Patients were informed about the study and their verbal and written informed consent was obtained. The study will be conducted in a public hospital in Istanbul with 68 patients (experimental group = 34, control group = 34) who met the research criteria and underwent CABG surgery. The patients in the experimental group will be given progressive relaxation exercises twice at 6-hour intervals on postoperative day 1 and day 2. Patients in the control group will receive routine treatment and care. Physiological parameters, pain, and anxiety levels will be evaluated twice daily on postoperative days 1 and 2 in both groups.It was also stated that a smart wristband should be worn on the arms of the patients on postoperative days 1 and 2 to monitor the frequency of mobilization in both the experimental and control groups. In addition, the frequency of analgesic use will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and write in Turkish,
* Analgesics given ≥4h before assessment,
* Conscious and communicative,
* Elective coronary artery bypass graft surgery planned,
* Patients undergoing coronary artery bypass graft surgery for the first time were included in the study.

Exclusion Criteria:

* Diagnosed with a psychiatric or neurological disorder,
* Diagnosis of a musculoskeletal condition that could affect mobilization,
* Patients with hearing and vision loss,
* Patients participating in another clinical trial during the same period,
* Patients who developed any complications during the postoperative period were excluded.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive Characteristics Form | Preoperative
  The first part includes questions about demographic characteristics such as gender, age, body mass index (height-weight), marital status, education level, income level and occupation, and the second part includes questions about other chronic diseases, previous surgery, previous stay in the intensive care unit, smoking and alcohol use.
Trait Anxiety Inventory | Preoperative
  The Trait Anxiety Inventory is used to determine how the individual "usually" feels and the items of the scale are scored between 1-4 points (1=almost never, 2=sometimes, 3=very often, 4=almost always). There are 7 reversed statements in the trait anxiety subscale (items 21, 26, 27, 30, 33, 36 and 39).
Physiological parameters monitoring | Postoperative Day 1:(measured twice, 6-hour apart): Control: Pre-test, 30 min later, 15 min post-mobilization Experimental: Pre-test, 5 min post-PGE, 15 min post-mobilization. Postoperative Day 2: Both groups:Same measurements at 6-hour intervals, twice
  Physiological parameters will be monitored.
State Anxiety Inventory | Postop Day 1:(measured twice, 6-hour apart): Control: Pre-test,30 minutes after,15 min post-mobilization.Experimental: Pre-test, 5 minutes after PGE, 15 min post-mobilization.Postoperative Day 2: Both groups:Same measurements at 6-hour intervals, twice
  It is used to determine how the individual feels "right now" and the items of the scale are scored between 1-4 points (1=not at all, 2=somewhat, 3=very much, 4=completely).
Short Form McGill Pain Questionnaire | Postop1:Measured twice at 6h:Control:Pre-test, 30 min later, post-mobilization vas, 15 min post-mobilization. Experimental: Pre-test, 5 min post-PGE, post-mobilization vas, 15 min post-mobilization.Postop2: Both groups:Measured twice at 6-hour intervals
  The scale consists of three parts in which the nature of pain, intensity of pain and overall pain intensity are evaluated.

SECONDARY OUTCOMES:
Mobilization Schedule | Postoperative day 1 and 2
  Mobilization will be assessed on postoperative days 1 and 2 based on the number of steps taken, distance covered, and relevant features of the mobilization process.
Analgesia monitoring form | Postoperative day 1 and 2
  In this form prepared by the researcher in line with the literature, the name, dose, time and route of administration will be recorded in case of analgesic use of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Koşuyolu Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the ethical approval for the study and the informed consent obtained from participants do not include permission to share data with third parties. Additionally, the responsibility to protect participant privacy and data confidentiality prevents such sharing.